CLINICAL TRIAL: NCT01291641
Title: Investigate Effect on Mean IMT of Probucol And/or CilosTazol in Patients With Coronary Heart dIsease Taking HMGCoA Reductase Inhibitor Therapy: A Randomized, Multicenter, Multinational Study
Brief Title: Effect of Probucol and/or Cilostazol on Mean IMT in Patients With Coronary Heart dIsease
Acronym: IMPACTonIMT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Byung-Hee Oh, Professor of Internal Medicine/Cardiology, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMT-01
Record Dates: First submitted 2011-01-31; First posted 2011-02-08 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Hyperlipidemias
Keywords: Hyperlipidemias; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Probucol; Cilostazol
MeSH Terms: conditions — Hyperlipidemias | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Probucol; Cilostazol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Placebo Comparator): HMGCoA reductase inhibitor continued
  Interventions: Drug: HMG-CoA Reductase Inhibitor
- Group B (Active Comparator): HMGCoA reductase inhibitor continued + Probucol 250 mg PO, BID
  Interventions: Drug: Probucol
- Group C (Active Comparator): HMGCoA reductase inhibitor continued + Probucol 250 mg PO, BID + Cilostazol 100 mg PO, BID
  Interventions: Drug: Cilostazol

INTERVENTIONS:
Drug: HMG-CoA Reductase Inhibitor — During the study period, HMGCoA reductase inhibitor is continuously administered to the patients.
  Dosage regimen: following the package insert of each HMGCoA reductase inhibitor
  Arms: Group A
Drug: Probucol — In addition to the continued HMGCoA reductase inhibitor treatment, probucol is administered.
  Dosage regimen: probucol 250-mg tablet, oral administration twice daily with meal(breakfast and dinner)
  Other Names: HMG-CoA Reductase Inhibitor
  Arms: Group B
Drug: Cilostazol — In addition to the continued HMGCoA reductase inhibitor treatment, probucol and cilostazol are administered.
  Dosage regimen: probucol 250-mg tablet, oral administration twice daily with meal(breakfast and dinner) Cilostazol 100-mg tablet, twice daily by the oral route
  Other Names: Probucol; HMG-CoA Reductase Inhibitor
  Arms: Group C

SUMMARY:
The purpose of this study is to evaluate the additional effect of probucol or concomitant administration of cilostazol and probucol on mean carotid artery intima-media thickness (mean IMT) at year 1, 2, and 3.

DETAILED DESCRIPTION:
Hyperlipidemic patients who are currently receiving HMGCoA reductase inhibitors(Statins) will be randomized Group A(Control), Group B(Probucol only added group) or Group C(Probucol and cilostazol added group) . Randomization will be done by the minimization method, controlling for the following factors: Country(Korea vs China) and max IMT (≥2.0mm vs.<2.0mm).

Group A : HMGCoA reductase inhibitor continued

Group B : HMGCoA reductase inhibitor continued + Probucol 250 mg PO, BID

Group C : HMGCoA reductase inhibitor continued + Probucol 250 mg PO, BID +Cilostazol 100 mg PO, BID

ELIGIBILITY:
Inclusion Criteria:

* 1) Subjects who are at least 20 y of age at the time of informed consent (male or female)
* 2) Subjects with coronary heart disease longer than 3 months.
* 3) Subjects being treated with HMGCoA reductase inhibitors(Statins)
* 4) Subjects with an max IMT equal to or greater than 1.2 mm
* 5) Subjects with an LDL-Cholesterol less than 200mg/dl
* 6) Subjects whose voluntary written informed consent is obtained for participation in this study

Exclusion Criteria:

* 1) Subjects who took probucol within 6 months before participation of the study
* 2) Subjects who took cilostazol within 3 months before participation of the study
* 3) Subjects with a history of hypersensitivity to probucol or cilostazol
* 4) Subjects with homozygous familial hyperlipidemia*
* 5) Subjects with a triglyceride ( TG) level greater than 400mg/dL at screening
* 6) Subjects with uncontrolled diabetes : HbA1c level greater than 9%
* 7) Subjects with New York Heart Association (NYHA) classification: Class Ⅲ and Ⅳ
* 8) Subjects with a QTc interval greater than 450msec(male) 470msec(female)
* 9) Subjects with serious ventricular arrythmias (frequent episodes of multifocal ventricular extrasystole)
* 10) Subjects with atrial fibrillation (including paroxysmal AF)
* 11) Subjects with unstable angina
* 12) Subjects with liver and kidney functions that satisfy the following criteria - AST or ALT >100 IU/L, serum creatinine >1.5 mg/dL
* 13) Subjects who are participating in another clinical trial
* 14) Subjects with pregnant or possibly pregnant without appropriate contraception control. Appropriate contraception control means that Oral contraception for greater than 4 weeks, surgical contraception including loop insertion, condom use etc. Women who has no possibility of pregnancy because of surgery or menopause should not be regarded the subject with possibly pregnant
* 15) Subjects with clinically significant disorders of blood coagulation
* 16) Subjects who are not considered by the physicians to be appropriate to participate in this trial for any other reason

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2011-03; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Difference of Carotid artery IMT (mean IMT) between screening and treatment completion(3 years after) or discontinuation | Baseline(screening), 3years
  For primary endpoint of Carotid artery IMT, t-test will be conducted for the mean IMT and variation by treatment arm(Group A vs B, Group A vs C). The 2-sided significance level is 5%. Morever, Mantel - Haenszel method can be accepted considering stratification factor or Sub-analysis can be done by each stratum in case of categorical variables.

SECONDARY OUTCOMES:
Time from enrollment date to the onset of composite cerebrovascular events | enrollment date, onset date(during study period, 3years)
  1. Cardiovascular death
  2. Myocardial infarction
  3. Cerebral infarction
  4. Unstable angina and cardiac failure, required hospitalization
  5. Coronary revascularization, required hospitalization
  6. PCI and coronary artery bypass grafting [CABG]
  Kaplan-Meier method will be conducted for the time from enrollment date to the onset of composite cerebrovascular and cardiovascular events by treatment arm(Group A vs B, Group A vs C). Overall survival curves and progression-free survival curves are estimated per treatment arm.
Number of composite cerebrovascular and cardiovascular events(including intervention) | enrollment date, onset date(during study period, 3years)
  1. Cardiovascular death
  2. Myocardial infarction
  3. Cerebral infarction
  4. Unstable angina and cardiac failure, required hospitalization
  5. Coronary revascularization, required hospitalization
  6. PCI and coronary artery bypass grafting [CABG]
  For the number of composite cerebrovascular and cardiovascular events (including intervention) t-test will be done by treatment arm(Group A vs B, Group A vs C).
The change of Biomarkers(1) | enrollment date ,onset date(during study period, 3years)
  Metabolic index: Lipid profile (TC, LDL-C, HDL-C, TG)
The change of Biomarkers(2) | enrollment date ,onset date(during study period, 3years)
  Inflammatory index: High sensitive C-reactive protein (hsCRP)
The change of Biomarkers(3) | enrollment date ,onset date(during study period, 3years)
  Oxidation index:oxidized LDL
  The change of biomarkers, t-test will be done by treatment arm(Group A vs B, Group A vs C).

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Hee Oh, M.D., Study Chair — Seoul National University Hospital; Cheol Ho Kim, M.D., Principal Investigator — Seoul National University Bundang Hospital; Sang-Hyun Kim, M.D., Principal Investigator — SMG-SNU Boramae Medical Center; Moo-Hyun Kim, M.D., Principal Investigator — Dong-A medical center
Locations (5):
- South Korea (5):
  - Dong-A Medical Center, Seogu, Busan
  - Samsung Medical Center, Seoul, Gangnam-Gu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Boramae Medical Center, Seoul

REFERENCES:
- [Result] Manzato E. Scandinavian simvastatin study (4S). Lancet. 1994 Dec 24-31;344(8939-8940):1767; author reply 1767-8. No abstract available. PMID 7997016
- [Result] Plehn JF, Davis BR, Sacks FM, Rouleau JL, Pfeffer MA, Bernstein V, Cuddy TE, Moye LA, Piller LB, Rutherford J, Simpson LM, Braunwald E. Reduction of stroke incidence after myocardial infarction with pravastatin: the Cholesterol and Recurrent Events (CARE) study. The Care Investigators. Circulation. 1999 Jan 19;99(2):216-23. doi: 10.1161/01.cir.99.2.216. PMID 9892586
- [Result] Long-Term Intervention with Pravastatin in Ischaemic Disease (LIPID) Study Group. Prevention of cardiovascular events and death with pravastatin in patients with coronary heart disease and a broad range of initial cholesterol levels. N Engl J Med. 1998 Nov 5;339(19):1349-57. doi: 10.1056/NEJM199811053391902. PMID 9841303
- [Result] Barnhart JW, Sefranka JA, McIntosh DD. Hypocholesterolemic effect of 4,4'-(isopropylidenedithio)-bis(2,6-di-t-butylphenol) (probucol). Am J Clin Nutr. 1970 Sep;23(9):1229-33. doi: 10.1093/ajcn/23.9.1229. No abstract available. PMID 5450842
- [Result] Tomikawa M, Nakayasu T, Tawara K, Abiko Y. Effect of probucol on serum lipoprotein levels in normal and dyslipoproteinemic mice. Atherosclerosis. 1981 Oct;40(2):101-13. doi: 10.1016/0021-9150(81)90029-0. PMID 6946776
- [Result] Tawara K, Tomikawa M, Abiko Y. Mode of action of probucol in reducing serum cholesterol in mice. Jpn J Pharmacol. 1986 Jan;40(1):123-33. doi: 10.1254/jjp.40.123. PMID 3959347
- [Result] Kita T, Nagano Y, Yokode M, Ishii K, Kume N, Ooshima A, Yoshida H, Kawai C. Probucol prevents the progression of atherosclerosis in Watanabe heritable hyperlipidemic rabbit, an animal model for familial hypercholesterolemia. Proc Natl Acad Sci U S A. 1987 Aug;84(16):5928-31. doi: 10.1073/pnas.84.16.5928. PMID 3475709
- [Result] Ishigami M, Yamashita S, Sakai N, Hirano K, Arai T, Maruyama T, Takami S, Koyama M, Kameda-Takemura K, Matsuzawa Y. High-density lipoproteins from probucol-treated patients have increased capacity to promote cholesterol efflux from mouse peritoneal macrophages loaded with acetylated low-density lipoproteins. Eur J Clin Invest. 1997 Apr;27(4):285-92. doi: 10.1046/j.1365-2362.1997.1040657.x. PMID 9134376
- [Result] Rinninger F, Wang N, Ramakrishnan R, Jiang XC, Tall AR. Probucol enhances selective uptake of HDL-associated cholesteryl esters in vitro by a scavenger receptor B-I-dependent mechanism. Arterioscler Thromb Vasc Biol. 1999 May;19(5):1325-32. doi: 10.1161/01.atv.19.5.1325. PMID 10323786
- [Result] Matsuzawa Y, Yamashita S, Funahashi T, Yamamoto A, Tarui S. Selective reduction of cholesterol in HDL2 fraction by probucol in familial hypercholesterolemia and hyperHDL2 cholesterolemia with abnormal cholesteryl ester transfer. Am J Cardiol. 1988 Jul 25;62(3):66B-72B. doi: 10.1016/s0002-9149(88)80055-9. PMID 3394656
- [Result] Daida H, Kuwabara Y, Yokoi H, Nishikawa H, Takatsu F, Nakata Y, Kutsumi Y, Oshima S, Nishiyama S, Ishiwata S, Kato K, Nishimura S, Miyauchi K, Kanoh T, Yamaguchi H. Effect of probucol on repeat revascularization rate after percutaneous transluminal coronary angioplasty (from the Probucol Angioplasty Restenosis Trial [PART]). Am J Cardiol. 2000 Sep 1;86(5):550-2, A9. doi: 10.1016/s0002-9149(00)01013-4. PMID 11009277
- [Result] Tardif JC, Cote G, Lesperance J, Bourassa M, Lambert J, Doucet S, Bilodeau L, Nattel S, de Guise P. Probucol and multivitamins in the prevention of restenosis after coronary angioplasty. Multivitamins and Probucol Study Group. N Engl J Med. 1997 Aug 7;337(6):365-72. doi: 10.1056/NEJM199708073370601. PMID 9241125
- [Result] Anderson TJ, Meredith IT, Yeung AC, Frei B, Selwyn AP, Ganz P. The effect of cholesterol-lowering and antioxidant therapy on endothelium-dependent coronary vasomotion. N Engl J Med. 1995 Feb 23;332(8):488-93. doi: 10.1056/NEJM199502233320802. PMID 7830729
- [Result] Sawayama Y, Shimizu C, Maeda N, Tatsukawa M, Kinukawa N, Koyanagi S, Kashiwagi S, Hayashi J. Effects of probucol and pravastatin on common carotid atherosclerosis in patients with asymptomatic hypercholesterolemia. Fukuoka Atherosclerosis Trial (FAST). J Am Coll Cardiol. 2002 Feb 20;39(4):610-6. doi: 10.1016/s0735-1097(01)01783-1. PMID 11849859
- [Result] Yamashita S, Bujo H, Arai H, Harada-Shiba M, Matsui S, Fukushima M, Saito Y, Kita T, Matsuzawa Y. Long-term probucol treatment prevents secondary cardiovascular events: a cohort study of patients with heterozygous familial hypercholesterolemia in Japan. J Atheroscler Thromb. 2008 Dec;15(6):292-303. doi: 10.5551/jat.e610. Epub 2008 Dec 6. PMID 19060422
- [Result] Bots ML, Grobbee DE. Intima media thickness as a surrogate marker for generalised atherosclerosis. Cardiovasc Drugs Ther. 2002 Jul;16(4):341-51. doi: 10.1023/a:1021738111273. PMID 12652104
- [Result] Crouse JR 3rd, Byington RP, Bond MG, Espeland MA, Craven TE, Sprinkle JW, McGovern ME, Furberg CD. Pravastatin, Lipids, and Atherosclerosis in the Carotid Arteries (PLAC-II). Am J Cardiol. 1995 Mar 1;75(7):455-9. doi: 10.1016/s0002-9149(99)80580-3. PMID 7863988
- [Result] de Groot E, Jukema JW, Montauban van Swijndregt AD, Zwinderman AH, Ackerstaff RG, van der Steen AF, Bom N, Lie KI, Bruschke AV. B-mode ultrasound assessment of pravastatin treatment effect on carotid and femoral artery walls and its correlations with coronary arteriographic findings: a report of the Regression Growth Evaluation Statin Study (REGRESS). J Am Coll Cardiol. 1998 Jun;31(7):1561-7. doi: 10.1016/s0735-1097(98)00170-3. PMID 9626835
- [Result] MacMahon S, Sharpe N, Gamble G, Hart H, Scott J, Simes J, White H. Effects of lowering average of below-average cholesterol levels on the progression of carotid atherosclerosis: results of the LIPID Atherosclerosis Substudy. LIPID Trial Research Group. Circulation. 1998 May 12;97(18):1784-90. doi: 10.1161/01.cir.97.18.1784. PMID 9603532
- [Result] Taylor AJ, Kent SM, Flaherty PJ, Coyle LC, Markwood TT, Vernalis MN. ARBITER: Arterial Biology for the Investigation of the Treatment Effects of Reducing Cholesterol: a randomized trial comparing the effects of atorvastatin and pravastatin on carotid intima medial thickness. Circulation. 2002 Oct 15;106(16):2055-60. doi: 10.1161/01.cir.0000034508.55617.65. PMID 12379573
- [Result] Baldassarre D, Franceschini G, Peruzzotti G, Brusoni B, Sirtori CR. Clinical evaluation of probucol in hypercholesteremia: individual lipoprotein responses and inhibitory effect on carotid atherosclerosis progression. J Cardiovasc Pharmacol. 1997 Dec;30(6):784-9. doi: 10.1097/00005344-199712000-00013. PMID 9436818
- [Result] Elam MB, Heckman J, Crouse JR, Hunninghake DB, Herd JA, Davidson M, Gordon IL, Bortey EB, Forbes WP. Effect of the novel antiplatelet agent cilostazol on plasma lipoproteins in patients with intermittent claudication. Arterioscler Thromb Vasc Biol. 1998 Dec;18(12):1942-7. doi: 10.1161/01.atv.18.12.1942. PMID 9848888
- [Result] Yoshikawa T, Mitani K, Kotosai K, Nozako M, Miyakoda G, Yabuuchi Y. Antiatherogenic effects of cilostazol and probucol alone, and in combination in low density lipoprotein receptor-deficient mice fed with a high fat diet. Horm Metab Res. 2008 Jul;40(7):473-8. doi: 10.1055/s-2008-1065348. Epub 2008 Apr 10. PMID 18404599
- [Result] Park SY, Lee JH, Shin HK, Kim CD, Lee WS, Rhim BY, Shin YW, Hong KW. Synergistic efficacy of concurrent treatment with cilostazol and probucol on the suppression of reactive oxygen species and inflammatory markers in cultured human coronary artery endothelial cells. Korean J Physiol Pharmacol. 2008 Aug;12(4):165-70. doi: 10.4196/kjpp.2008.12.4.165. Epub 2008 Aug 31. PMID 19967051
- [Result] Smilde TJ, van Wissen S, Wollersheim H, Trip MD, Kastelein JJ, Stalenhoef AF. Effect of aggressive versus conventional lipid lowering on atherosclerosis progression in familial hypercholesterolaemia (ASAP): a prospective, randomised, double-blind trial. Lancet. 2001 Feb 24;357(9256):577-81. doi: 10.1016/s0140-6736(00)04053-8. PMID 11558482